CLINICAL TRIAL: NCT02000778
Title: A Pilot & Feasibility Study of the Imaging Potential of EC17 in Subjects Undergoing Intraoperative Detection of Occult Ovarian Carcinoma
Brief Title: EC17 for Intraoperative Imaging in Occult Ovarian Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 818533; 818533 [UPenn IRB Protocol #]
Record Dates: First submitted 2013-11-26; First posted 2013-12-04 (Estimated); Last update posted 2018-06-04 (Actual); Status verified 2017-03

CONDITIONS: Ovarian Cancer
Keywords: Occult Ovarian Carcinoma
MeSH Terms: conditions — Ovarian Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- EC17 Injection Group (Experimental): The group will receive a single dose of EC17, infused over 10 minutes, prior to surgery. Then, during surgery, the EC-17 will be imaged with a camera that the investigators have developed.
  Interventions: Drug: EC17

INTERVENTIONS:
Drug: EC17
  Other Names: Folate-FITC

SUMMARY:
The overall prevalence of Ovarian Cancer in the United States according to the US SEER Registry is 182,710 women. Ovarian cancer also has the highest mortality rate of the gynecological cancers. The overall five-year survival rate is 45% and for Stages III and IV it is only 20-25%. The majority of these are aged 50 years or older, but a few girls less than 10 years of age have been diagnosed with ovarian cancer. This risk increases with age and decreases with numbers of pregnancies.

The prognosis for many carcinomas is dependent on the extent of surgical resection. At present, the ability to perform a complete resection with negative margins is limited by the investigator's ability to palpate and visualize the tumor and its borders. In many cases, a more radical resection than necessary is performed in order to provide assurance that negative margins are achieved. This approach may also increase complication rates, as well as short- and long-term morbidity. It is desirable to improve visualization of primary tumors and occult metastases in real time, during surgery. The use of fluorescent probes that recognize cancer-specific antigens, in conjunction with a clinical imaging system, is under investigation.

Ovarian cancer is a prototypic disease for this type of clinical imaging system called intra-operative imaging. Except in Stage IV, the tumors are confined to the pelvis or abdomen and typically involve extensions or implants onto pelvic or abdominal organs or membranes. Tumor debulking surgery is common early in the disease process as many of the tumors can be identified by appearance or feel in the skilled surgeon's hands. The major problems are that tumors can be diffuse and numerous, of various sizes, and often not readily visible in the surgical field.

Over 90-95% of serous ovarian cancers express folate receptor (FR)-alpha, making this receptor an ideal target for marking most ovarian cancers. Folate is the prototypic agonist at the FR-alpha with potential uses for imaging and targeted therapeutic strategies.Chemotherapy does not affect FR-alpha expression in ovarian cancer specimens examined by immunohistochemistry, so prior treatment is unlikely to affect utility of FR-alpha agonists as imaging or therapeutic agents.

ELIGIBILITY:
Inclusion Criteria:

1. Female subjects 18 years of age and older
2. Female subjects of childbearing potential or less than 2 years postmenopausal agree to receive a urinary or serum beta HCG test prior to subject enrollment. Documentation must be acquired for women of menopausal or post-menopausal status prior to subject enrollment if they are below the age of sixty (60).
3. Primary diagnosis, or at high clinical suspicion, of primary ovarian cancer:

   1. Patient is scheduled to undergo laparotomy OR
   2. Patient is scheduled to undergo laparoscopy then pre-authorized laparotomy if cancer is found.

Exclusion Criteria:

1. Known sarcomatous histologies

1. Recurrent ovarian cancer
2. Known FR-alpha negative cancer
3. Planned surgical approach via laparoscopy or robotic (no intention to perform laparotomy)
4. History of anaphylactic reactions to Folate-FITC (EC17) or insects
5. Pregnancy
6. Brain metastases
7. Taking compounds that inhibit active transport of organic anions (probenecid)
8. Hepatic impairment, as evidenced by greater than 3x the upper limit of normal (ULN) for ALT, AST, or total bilirubin (except for known cases of Gilbert's syndrome), or renal impairment, as evidenced by greater than 1.5x the ULN for BUN or creatinine
9. Received study agent in another investigational drug or vaccine trial prior to surgery
10. At-risk patient populations

    1. People who would easily be lost to follow up (ex: People who are homeless or alcohol dependent)
    2. Patients unable to participate in the consent process (children and neonates)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2013-11; Primary Completion 2014-11-12 (Actual); Study Completion 2014-11-12 (Actual)

PRIMARY OUTCOMES:
The ability of EC17 and the imaging system to detect FRA positive tumors during surgery conducted 2-4 hours post EC-17 administration. | Within two to four hours of injection of EC17

SECONDARY OUTCOMES:
The number of participants that will have an adverse reaction to the EC17 | Day 1-Day 30

CONTACTS AND LOCATIONS:
Overall Officials: Sunil Singhal, Principal Investigator — University of Pennsylvania
Locations (1):
- Hospital of the University of Pennsylvania, Philadelphia, Pennsylvania, United States